CLINICAL TRIAL: NCT00930462
Title: A Prospective Randomised Controlled Trial Comparing Cap-Assisted Colonoscopy Versus Standard Colonoscopy
Brief Title: Evaluation of the Use of Cap in Improving the Performance of Colonoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Royal Prince Alfred Hospital, Sydney, Australia (Other)
Responsible Party: Hoi-Poh Tee, Royal Prince Alfred Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CAPCOLON; X07-0107
Record Dates: First submitted 2009-06-26; First posted 2009-06-30 (Estimated); Last update posted 2009-06-30 (Estimated); Status verified 2009-06

CONDITIONS: Colonoscopy
Keywords: colonoscopy; cap; hood; cecal intubation time; polyp detection rate; performance
MeSH Terms: conditions — Anterior polar cataract 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional colonoscopy (No Intervention): No cap fitted on the colonoscopes for this group.
- Cap-assisted colonoscopy (Experimental)
  Interventions: Device: Cap (Olympus Medical Systems: D-201-15004, D-201-14304 and D-201-12704)

INTERVENTIONS:
Device: Cap (Olympus Medical Systems: D-201-15004, D-201-14304 and D-201-12704) — Plastic cap fitted on the colonoscope
  Other Names: D-201-15004, D-201-14304 and D-201-12704; Olympus Medical Systems, Tokyo, Japan.
  Arms: Cap-assisted colonoscopy

SUMMARY:
The aim of this study is to compare the colonoscopy success rate, cecal time and polyp detection rate between cap-fitted colonoscopy and conventional colonoscopy.

DETAILED DESCRIPTION:
Colonoscopic examination has been used in clinical practice for approximately 40 years. Despite the fact that colonoscopy is widely available and is performed by many experienced colonoscopists there are concerns about the quality of colonoscopy as measured by several technical endpoints such as rate of failed caecal intubation and polyp miss rate. A large population-based study revealed 13.1% of colonoscopies failed to reach the cecum. In addition, one large review of back-to-back colonoscopies showed polyp miss rates of 24% for adenoma.

One potentially promising technique is cap-assisted colonoscopy. A transparent cap (or "hood") is a simple plastic device that can be attached to the tip of a colonoscope before performing the colonoscopy. Several randomized trials from Japan have mixed results regarding improved cecal intubation times and polyp detection rates. A recent large study from Hong Kong showed improved time to cecum but a reduced polyp detection rate. To date there is no large randomized study using the cap in a western population, in whom the colorectal cancer (CRC) incidence is known to be higher. We plan to conduct a randomized controlled trial to investigate the usefulness of cap-assisted colonoscopy in a Western population.

ELIGIBILITY:
Inclusion Criteria:

* All colonoscopy patients referred for colonoscopy at Royal Prince Alfred Hospital.

Exclusion Criteria:

* Prior colonic resection
* Pregnancy.
* Severe co-morbidities.
* Tertiary referral for endo-mucosal resection.
* Acute surgical conditions such as severe colitis, toxic megacolon, ischemic colitis, acute gastrointestinal bleeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2008-03; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Time to cecum | One month

SECONDARY OUTCOMES:
Polyp detection rate | One month

CONTACTS AND LOCATIONS:
Overall Officials: Arthur J Kaffes, FRACP, Principal Investigator — Royal Prince Alfred Hospital, Sydney
Locations (1):
- Royal Prince Alfred Hospital, Sydney, New South Wales, Australia

REFERENCES:
- [Result] Lee YT, Lai LH, Hui AJ, Wong VW, Ching JY, Wong GL, Wu JC, Chan HL, Leung WK, Lau JY, Sung JJ, Chan FK. Efficacy of cap-assisted colonoscopy in comparison with regular colonoscopy: a randomized controlled trial. Am J Gastroenterol. 2009 Jan;104(1):41-6. doi: 10.1038/ajg.2008.56. PMID 19098847
- [Result] Kondo S, Yamaji Y, Watabe H, Yamada A, Sugimoto T, Ohta M, Ogura K, Okamoto M, Yoshida H, Kawabe T, Omata M. A randomized controlled trial evaluating the usefulness of a transparent hood attached to the tip of the colonoscope. Am J Gastroenterol. 2007 Jan;102(1):75-81. doi: 10.1111/j.1572-0241.2006.00897.x. Epub 2006 Nov 13. PMID 17100978
- [Result] Harada Y, Hirasawa D, Fujita N, Noda Y, Kobayashi G, Ishida K, Yonechi M, Ito K, Suzuki T, Sugawara T, Horaguchi J, Takasawa O, Obana T, Oohira T, Onochi K, Kanno Y, Kuroha M, Iwai W. Impact of a transparent hood on the performance of total colonoscopy: a randomized controlled trial. Gastrointest Endosc. 2009 Mar;69(3 Pt 2):637-44. doi: 10.1016/j.gie.2008.08.029. PMID 19251004
- [Result] Shida T, Katsuura Y, Teramoto O, Kaiho M, Takano S, Yoshidome H, Miyazaki M. Transparent hood attached to the colonoscope: does it really work for all types of colonoscopes? Surg Endosc. 2008 Dec;22(12):2654-8. doi: 10.1007/s00464-008-9790-6. Epub 2008 Feb 23. PMID 18297353
- [Derived] Tee HP, Corte C, Al-Ghamdi H, Prakoso E, Darke J, Chettiar R, Rahman W, Davison S, Griffin SP, Selby WS, Kaffes AJ. Prospective randomized controlled trial evaluating cap-assisted colonoscopy vs standard colonoscopy. World J Gastroenterol. 2010 Aug 21;16(31):3905-10. doi: 10.3748/wjg.v16.i31.3905. PMID 20712051